CLINICAL TRIAL: NCT03720769
Title: Increasing Access to Mental Health Care for People Living in Lebanon: An E-Mental Health Intervention
Brief Title: Testing e-Mental Health in Lebanon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VU University of Amsterdam (Other)
Collaborators: World Health Organization (Other); Ministry of Public Health, Lebanon (Unknown); Freie Universität Berlin (Other)
Responsible Party: Principal Investigator, Pim Cuijpers, Professor, VU University of Amsterdam
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERC.0002797
Record Dates: First submitted 2018-10-24; First posted 2018-10-25 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Step-by-Step (Experimental)
  Interventions: Behavioral: Step-by-Step
- Enhanced care as usual (Active Comparator)
  Interventions: Behavioral: Enhanced care as usual

INTERVENTIONS:
Behavioral: Step-by-Step — Guided self-help programme delivered through an app/website for the treatment of depression
  Arms: Step-by-Step
Behavioral: Enhanced care as usual — Psychoeducation and information about where to get help (i.e., mhGAP trained primary health care centres)
  Arms: Enhanced care as usual

SUMMARY:
The study objective is to test a guided e-mental health intervention called Step-by-Step for people living in Lebanon. Step-by-Step is a self-help programme delivered through an app or website and aims to treat symptoms of depression and other symptoms of psychological distress. First, a small study will be conducted to test the research procedure. Second, a large study will be conducted to test the effectiveness of Step-by-Step.

People residing in Lebanon (i.e. Lebanese, Palestinians and Syrian displaced people), above the age of 18 with symptoms of depression will be recruited through social media, posters, radio and television adverts, etc. Minors (under the age of 18) and people who have plans to end their life will be excluded from the study.

To test whether the use of Step-by-Step improves symptoms of depression, two groups will be compared. Participants in the intervention group will receive Step-by-Step, while those in the control group will receive basic information about depression and a list of health centres where they can get face-to-face help that is based on evidence. In addition, participants in the intervention group will receive weekly phone or chat support (up to 15 minutes) provided through lay helpers who were trained and work under the supervision of a trained clinical psychologist. The study hypothesises that participants who receive Step-by-Step will have a higher symptom improvement than participants who receive basic information.

In order to assess symptoms of depression and other symptoms of psychological distress, participants in this study will complete several questionnaires three times: At the beginning of the study, after 8 weeks, and then three months later (i.e. 5 months after the beginning of the study).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or above
* PHQ-9 sum score above 9
* WHODAS 2.0 sum score above 16

Exclusion Criteria:

* Serious thoughts or plans to end one's life

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1248 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2020-09-16 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | 8 weeks
  Self-administered instrument for depression screening (intention-to-treat analysis)
WHO Disability Assessment Schedule 2.0 (WHODAS 2.0) | 8 weeks
  Generic assessment instrument for health and disability (intention-to-treat analysis)

SECONDARY OUTCOMES:
WHO-5 Well-Being Index | 8 weeks
Generalized Anxiety Disorder - 7 Questionnaire (GAD-7) | 8 weeks
PTSD Checklist for DSM-5 (PCL-6) | 8 weeks
Self-defined psychosocial problems (PSYCHLOPS) | 8 weeks
(Adapted) Client Service Receipt Inventory (CSRI) | 8 weeks

OTHER OUTCOMES:
Client Satisfaction Questionnaire (CSQ-3) | only at post-assessment (8 weeks after baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Pim Cuijpers, Professor, Principal Investigator — VU Amsterdam
Locations (1):
- Ministry of Public Health, Beirut, Lebanon

REFERENCES:
- [Derived] Abi Ramia J, Khoury S, Armani N, Cuijpers P, Carswell K, van 't Hof E, Zoghbi E, Sijbrandij M, El Chammay R. From research to real-life implementation: an evaluation of the scale up of a guided digital mental health intervention in Lebanon: Step-by-Step. Front Public Health. 2025 Nov 11;13:1665093. doi: 10.3389/fpubh.2025.1665093. eCollection 2025. PMID 41306862
- [Derived] Abi Hana R, Abi Ramia J, Burchert S, Carswell K, Cuijpers P, Heim E, Knaevelsrud C, Noun P, Sijbrandij M, van Ommeren M, Van't Hof E, Wijnen B, Zoghbi E, El Chammay R, Smit F. Cost-Effectiveness of Digital Mental Health Versus Usual Care During Humanitarian Crises in Lebanon: Pragmatic Randomized Trial. JMIR Ment Health. 2024 May 29;11:e55544. doi: 10.2196/55544. PMID 38810255
- [Derived] Cuijpers P, Heim E, Abi Ramia J, Burchert S, Carswell K, Cornelisz I, Knaevelsrud C, Noun P, van Klaveren C, Van't Hof E, Zoghbi E, van Ommeren M, El Chammay R. Effects of a WHO-guided digital health intervention for depression in Syrian refugees in Lebanon: A randomized controlled trial. PLoS Med. 2022 Jun 23;19(6):e1004025. doi: 10.1371/journal.pmed.1004025. eCollection 2022 Jun. PMID 35737665
- [Derived] Cuijpers P, Heim E, Ramia JA, Burchert S, Carswell K, Cornelisz I, Knaevelsrud C, Noun P, van Klaveren C, Van't Hof E, Zoghbi E, van Ommeren M, El Chammay R. Guided digital health intervention for depression in Lebanon: randomised trial. Evid Based Ment Health. 2022 Dec;25(e1):e34-e40. doi: 10.1136/ebmental-2021-300416. Epub 2022 May 16. PMID 35577536
- [Derived] van 't Hof E, Heim E, Abi Ramia J, Burchert S, Cornelisz I, Cuijpers P, El Chammay R, Harper Shehadeh M, Noun P, Smit F, van Klaveren C, van Ommeren M, Zoghbi E, Carswell K. Evaluating the Effectiveness of an E-Mental Health Intervention for People Living in Lebanon: Protocol for Two Randomized Controlled Trials. JMIR Res Protoc. 2021 Jan 28;10(1):e21585. doi: 10.2196/21585. PMID 33507158